CLINICAL TRIAL: NCT03545139
Title: Clinical and Radiographic Evaluation of Neo MTA Versus Conventional White MTA in Revascularization of Non-Vital Immature Permanent Anterior Teeth: A Randomized Controlled Trial
Brief Title: Clinical & Radiographic Evaluation of Neo MTA Versus White MTA in Revascularization of Non-Vital Immature Permanent Teeth
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Ahmed Tawfik, Researcher assistant at orthodontic and pediatric dentistry department National Research centre, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeoMTA in Revascularization
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Nonvital Tooth
Keywords: pulp revascularization; endodontic regeneration; NeoMTA
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NeoMTA (intervention group) (Experimental): Revascularization with NeoMTA as coronal plug.
  Interventions: Biological: NeoMTA nusmile
- White MTA (Control group) (Active Comparator): Revascularization with Conventional white mineral trioxide aggregate (White MTA) as coronal plug.
  Interventions: Biological: White MTA

INTERVENTIONS:
Biological: NeoMTA nusmile — A new formulation of MTA was developed in which bismuth oxide was omitted.
  Arms: NeoMTA (intervention group)
Biological: White MTA — Revascularization with Conventional white mineral trioxide aggregate as coronal plug.
  Arms: White MTA (Control group)

SUMMARY:
* To evaluate and compare the degree of tooth discoloration in tooth crowns induced by Neo MTA versus white MTA over time.
* Evaluation of the effectiveness of Neo MTA as coronal plug in revascularization of immature teeth with necrotic pulp.

DETAILED DESCRIPTION:
The new formulation of MTA (NeoMTA) does not contain bismuth oxide, will be used in revascularization of nonvital immature permanent anterior teeth.

to evaluate the effectiveness of Neo MTA as coronal plug and compare the degree of tooth discoloration in tooth crowns induced by Neo MTA versus white MTA over time.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients: 7-15years old.
* Free from any systemic diseases that may affect the normal healing process.
* Tooth with immature root apex.
* Traumatically or cariously exposed non vital permanent anterior tooth.
* Pulp space not needed for post and core for final restoration.
* Compliant patient/parent

Exclusion Criteria:

* Patients having allergy to medicaments and antibiotics necessary to complete procedure.
* Tooth with vital pulp or complete root formation.
* Teeth with internal or external root resorption.
* Un-cooperative patients.
* Luxative injuries.
* Teeth with a root fracture
* Alveolar fracture
* Subjects with chronic systemic illness.
* Subjects with poor oral hygiene.
* Compromised remaining tooth structure as teeth with extensive loss of coronal tissue will require restoration with a post that will occupy the space required for blood clot formation.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Discoloration/ Staining potential | 9 month
  Using spectrophotometer by operator

SECONDARY OUTCOMES:
Pain on biting | 9 month
  Verbal questioning of the patient
Pain on percussion | 9 month
  Using back of the mirror
Sinus or fistula, recurrent swelling | 9 month
  Visual examination by operator
Root lengthening | 9 month
  Radiographic Digora image analysis software i.e. Digora for windows software DFW

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral & Dental Medicine Cairo University, Cairo, Egypt